CLINICAL TRIAL: NCT07374328
Title: Comparison Of Two Triple Hypoglycemic Regimens In Achieving Glycemic Control And Diabetes Remission In Hospitalized Patients With Newly Diagnosed Type 2 Diabetes Mellitus: A Multicenter, Randomized, Clinical Study
Brief Title: Triple Hypoglycemic Regimens In Patients With Newly Diagnosed Type 2 Diabetes Mellitus
Acronym: TRED
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRED
Record Dates: First submitted 2025-12-11; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: triple regimen; diabetes; remission
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — semaglutide; Sitagliptin Phosphate; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide group: patients receive semaglutide treatment. (Experimental): Patients receive 0.25 mg per week in the first month, 0.5 mg per week in the second month, and 1.0mg of semaglutide per week from the 3rd to the 8th month.
  Interventions: Drug: Semaglutide (1 Mg Dose)
- Oral medication group: patients receive triple hypoglycemic oral medications. (Active Comparator): Patients in oral medication group received sitagliptin 0.1g per day. Both groups were simultaneously treated with metformin (1.0g daily, divided into two doses) and empagliflozin (10mg daily).
  Interventions: Drug: Sitagliptin (DPP4 inhibitor)

INTERVENTIONS:
Drug: Semaglutide (1 Mg Dose) — 0.25 mg per week in the first month, 0.5 mg per week in the second month, and 1.0mg of semaglutide per week from the 3rd to the 8th month.
  Arms: Semaglutide group: patients receive semaglutide treatment.
Drug: Sitagliptin (DPP4 inhibitor) — Sitagliptin 0.1g per day.
  Arms: Oral medication group: patients receive triple hypoglycemic oral medications.

SUMMARY:
This study is a multicenter, randomized, controlled study. A sample size of 240 cases is proposed to be included. The inclusion criteria are: (1) patients with newly diagnosed type 2 diabetes; (2) age between 18 and 65 years old; (3) HbA1c ≥ 9.0%. The exclusion criteria include: (1) type 1 diabetes; (2) elevated creatinine or urinary albumin/creatinine; (3) combined with coronary heart disease, tumor or pregnancy; (4) receiving glucocorticoids. The selected participants are randomly divided into two groups: one group is the semaglutide group, and the other isthe oral medication group. The treatment plan is as follows. Semaglutide group: 0.25 mg per week in the first month, 0.5 mg per week in the second month, and 1.0mg per week from the 3rd to the 8th month of semaglutide. Oral medication group: Sitagliptin 0.1g per day. Both groups were simultaneously treated with metformin (1.0g daily, divided into two doses) and empagliflozin (10mg daily). The first phase of the study was as follows: Semaglutide group: Treatment was initiated until 6 months after the titration dose of 1mg was reached; Oral medication group: Initiate treatment until 6 months after reaching a fixed dose. At the end of the first stage of the study, for the selected participants with HbA1c<6.5%, the hypoglycemic drugs were discontinued and they entered the second stage of the study. The study was concluded after a 3-month follow-up. The evaluation indicators include: effectiveness indicators (HbA1c, diabetes remission rate, continuous glucose monitoring), safety indicators (hypoglycemia, adverse reactions, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed type 2 diabetes.
* Age between 18 and 65 years old.
* HbA1c ≥ 9.0%.

Exclusion Criteria:

* Type 1 diabetes.
* Elevated creatinine or urinary albumin/creatinine.
* Combined with coronary heart disease, tumor or pregnancy.
* Receiving glucocorticoids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes remission rate | From enrollment to the end of follow-up at 11 months

SECONDARY OUTCOMES:
HbA1c | From enrollment to the end of follow-up at 11 months
Hypoglycemia rate | From enrollment to the end of follow-up at 11 months
Adverse reactions | From enrollment to the end of follow-up at 11 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Guangzhou Medical University, Guangzhou, Guangdong, China